CLINICAL TRIAL: NCT01283490
Title: The Effect of Sonophoresis on Topical Anesthesia: a Clinical Trial
Brief Title: The Effect of Sonophoresis on Topical Anesthesia: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Innovadontics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 5100300
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Topical Anesthetic Applied With Sonophoresis
Keywords: topical anesthetic, sonophoresis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DASD Group (Active Comparator): Benzocaine 20% will be placed using the DASD for one minute. Immediately after DASD application a needle puncture with a 27 gauge needle to the depth of 3 millimeters will be performed.
  Interventions: Device: DASD Group
- Sonic Vibration (SV) (Sham Comparator): A modified tooth brush which only allows sonic vibration (SV), that has the appearance and sound of the DASD will be used to apply the benzocaine 20% for one minute. Following application with the SV a needle puncture with a 27 gauge needle to the depth of 3millimeters.
  Interventions: Device: Sonic Vibration (SV)

INTERVENTIONS:
Device: DASD Group — Single application of 20% Benzocaine applied for one minute with the DASD ultrasonic and sonic vibration prior to needle puncture.
  Arms: DASD Group
Device: Sonic Vibration (SV) — Single application of 20% benzocaine applied with SV for one minute prior to needle puncture.
  Arms: Sonic Vibration (SV)

SUMMARY:
The Dental Anesthesia Sonophoresis Device (DASD) is a novel device that is intended to reduce the discomfort associated with puncturing the oral mucosa. DASD is a portable, battery-powered device that simultaneously generates ultrasonic energy and sonic vibration in a small applicator head that can easily reach and adapt to injection sites in the oral cavity. The ultrasonic energy provides a sonophoretic effect on the oral mucosa, generating micro channels through the lipids between the keratinized cells that make up the stratum corneum. Once the benzocaine has permeated the stratum corneum, it is quickly absorbed into the soft tissue desensitizing the area and reducing the perception of pain caused by the trauma of puncturing soft tissue. Methods: A split-mouth model using 50 healthy subjects from the ages of 18 to 50 will undergo needle puncture of the maxillary mucobuccal fold at the canine eminence. Prior to the injection there will be randomized application of 20% Benzocaine with a device which is a modified battery operated tooth brush that in appearance and sound is similar to the DASD which only produces sonic vibration which will be known as (SV) or 20% benzocaine with application of the DASD device, that produces ultrasonic as well as sonic vibration. Subjects will rate their pain according to the Visual Analog Scale (VAS).The purpose of this study is to evaluate whether sonophoresis applied using the DASD will eliminate the pain associated with intraoral injections within one minute of application.

Null Hypothesis (Ho): There is no difference in the perception of pain when the DASD is used compared to topical anesthetic applied with sonic vibration.

The Alternative Hypothesis (Ha): There is a difference in pain perception when the DASD is used for application of topical anesthetic compared to topical anesthetic applied with sonic vibration.

DETAILED DESCRIPTION:
Fifty healthy patients between the ages of 18 and 50 will be used for this clinical trial. The anatomical site used for this clinical trial is the maxillary mucobuccal fold above the canine eminence. This site has been selected because it is an anatomical structure that is easily found for all subjects and is reproducible from one side of the patient to the other. One side of the patient's maxillary mucobuccal canine area will be dried with dental 2x2 sponge gauze, then 20% Benzocaine will be applied with an SV for one minute. The site will then be punctured using a short 27-gauge needle inserted to the depth of 3mm.

Immediately after the removal of the needle, the patients will be asked to rate their pain according to the Visual Analogue Scale (VAS) model. The VAS is a measurement instrument 100mm in length anchored by word descriptors at each end. The subject marks on the line the point that they feel represents their perception of their current state.

On the contralateral side, a 2x2 will be used to dry the mucus, and then 20% benzocaine will be applied using the DASD for one minute, followed by a puncture of the oral mucosa with a 27-gauge needle to the depth of 3mm. Immediately after the removal of the needle, the subject will rate their pain according to the same method described above. The application of the topical anesthetic by the DASD and SV will be administered by a single investigator for all subjects. After administration of topical anesthetic the subjects will be divided randomly among six separate investigators who will insert the needle into the mucosa. Neither the investigator giving the injection nor the subjects will be told whether the DASD or SV was used to administer the topical anesthesia. This will insure a double blind trial. A new 27-gauge needle will be used for each injection site to standardize each injection.

Statistical Analysis

Each patient will be treated prior to injection with a topical anesthetic applied either using the SV device or the DASD device. A paired t-test will be used to determine if a statistically significant difference exists between pain scores recorded for each of the injection sites. For the VAS model, the patient's vertical mark is measured from the left hand side in millimeters. The paired t-test will test if the mean difference between SV treated sites and DASD, treated sites to determine which of the two hypotheses are true. The Null Hypothesis (Ho) is that the mean of the differences in pain scores is zero. The Alternative Hypothesis (Ha) is that the mean of the differences in pain scores is not equal to zero . A probability value of 0.05 will be used to determine if the difference is significant.

ELIGIBILITY:
Inclusion Criteria:

1. Good general health as evidenced by the medical history.
2. Ages 18 to 50 (male or female).

Exclusion Criteria:

1. Use of tobacco products.
2. A soft or hard tissue tumor of the oral cavity.
3. Advanced periodontal disease (characterized by the presence of purulent exudate, tooth mobility, and/or extensive alveolar bone loss).
4. Participation in another clinical study or panel test.
5. Pregnant women or women who are breast-feeding.
6. Diabetic.
7. Allergy to benzocaine or ester-type local anesthetic.
8. Previous dental treat in experimental area within 30 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The Effect of Sonophoresis on Topical Anesthesia: a Clinical Trial | Immediately after needle puncture
  Subjects will rate there perceived pain immediately after needle puncture using the Visual Analog Scale (VAS). This will occur twice once after application of topical anesthetic by a dummy device and another after application of topical anesthetic with the Dental Anesthesia Sonophoresis Device (DASD)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Torabinejad, DMD MSD PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

REFERENCES:
- [Background] Calatayud J, Gonzalez A. History of the development and evolution of local anesthesia since the coca leaf. Anesthesiology. 2003 Jun;98(6):1503-8. doi: 10.1097/00000542-200306000-00031. No abstract available. PMID 12766665
- [Background] Giddon DB, Quadland M, Rachwall PC, Springer J, Tursky B. Development of a method for comparing topical anesthetics in different application and dosage forms. J Oral Ther Pharmacol. 1968 Jan;4(4):270-4. No abstract available. PMID 4868310
- [Background] Carr MP, Horton JE. Clinical evaluation and comparison of 2 topical anesthetics for pain caused by needle sticks and scaling and root planing. J Periodontol. 2001 Apr;72(4):479-84. doi: 10.1902/jop.2001.72.4.479. PMID 11338300
- [Background] Martin MD, Ramsay DS, Whitney C, Fiset L, Weinstein P. Topical anesthesia: differentiating the pharmacological and psychological contributions to efficacy. Anesth Prog. 1994;41(2):40-7. PMID 8638859
- [Background] Fukayama H, Suzuki N, Umino M. Comparison of topical anesthesia of 20% benzocaine and 60% lidocaine gel. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2002 Aug;94(2):157-61. doi: 10.1067/moe.2002.124858. PMID 12221381
- [Background] Nakanishi O, Haas D, Ishikawa T, Kameyama S, Nishi M. Efficacy of mandibular topical anesthesia varies with the site of administration. Anesth Prog. 1996 Winter;43(1):14-9. PMID 10323120
- [Background] Hutchins HS Jr, Young FA, Lackland DT, Fishburne CP. The effectiveness of topical anesthesia and vibration in alleviating the pain of oral injections. Anesth Prog. 1997 Summer;44(3):87-9. PMID 9481967
- [Background] Vickers ER, Punnia-Moorthy A. A clinical evaluation of three topical anaesthetic agents. Aust Dent J. 1992 Aug;37(4):267-70. PMID 1444945
- [Background] Rosivack RG, Koenigsberg SR, Maxwell KC. An analysis of the effectiveness of two topical anesthetics. Anesth Prog. 1990 Nov-Dec;37(6):290-2. PMID 2097909
- [Background] Chung JE, Koh SA, Kim TI, Seol YJ, Lee YM, Ku Y, Rhyu IC, Chung CP, Koo KT. Effect of eutectic mixture of local anesthetics on pain perception during scaling by ultrasonic or hand instruments: a masked randomized controlled trial. J Periodontol. 2011 Feb;82(2):259-66. doi: 10.1902/jop.2010.090748. Epub 2010 Aug 23. PMID 20731585
- [Background] Musawi AA, Andersson L. Use of topical as only anesthetic for suturing a traumatic facial laceration. Dent Traumatol. 2010 Jun;26(3):292-3. doi: 10.1111/j.1600-9657.2010.00881.x. PMID 20572847
- [Background] Meechan JG. Intra-oral topical anaesthetics: a review. J Dent. 2000 Jan;28(1):3-14. doi: 10.1016/s0300-5712(99)00041-x. PMID 10666956
- [Background] Meechan JG. Effective topical anesthetic agents and techniques. Dent Clin North Am. 2002 Oct;46(4):759-66. doi: 10.1016/s0011-8532(02)00035-6. PMID 12436830
- [Background] Watanabe IS. Ultrastructures of mechanoreceptors in the oral mucosa. Anat Sci Int. 2004 Jun;79(2):55-61. doi: 10.1111/j.1447-073x.2004.00067.x. PMID 15218624
- [Background] Swartzendruber DC. Studies of epidermal lipids using electron microscopy. Semin Dermatol. 1992 Jun;11(2):157-61. PMID 1498019
- [Background] Squier CA. The permeability of keratinized and nonkeratinized oral epithelium to horseradish peroxidase. J Ultrastruct Res. 1973 Apr;43(1):160-77. doi: 10.1016/s0022-5320(73)90076-2. No abstract available. PMID 4703271
- [Background] Gangarosa LP Sr. Newer local anesthetics and techniques for administration. J Dent Res. 1981 Aug;60(8):1471-80. doi: 10.1177/00220345810600080906. No abstract available. PMID 6942011
- [Background] Malamed SF. What's new in local anesthesia? Anesth Prog. 1992;39(4-5):125-31. No abstract available. PMID 1344014
- [Background] Mitragotri S, Kost J. Low-frequency sonophoresis: a review. Adv Drug Deliv Rev. 2004 Mar 27;56(5):589-601. doi: 10.1016/j.addr.2003.10.024. PMID 15019748
- [Background] Benson HA, McElnay JC, Harland R, Hadgraft J. Influence of ultrasound on the percutaneous absorption of nicotinate esters. Pharm Res. 1991 Feb;8(2):204-9. doi: 10.1023/a:1015892020468. PMID 2023868
- [Background] Tachibana K, Tachibana S. Use of ultrasound to enhance the local anesthetic effect of topically applied aqueous lidocaine. Anesthesiology. 1993 Jun;78(6):1091-6. doi: 10.1097/00000542-199306000-00011. PMID 8512102
- [Background] Mitragotri S, Blankschtein D, Langer R. Ultrasound-mediated transdermal protein delivery. Science. 1995 Aug 11;269(5225):850-3. doi: 10.1126/science.7638603.